CLINICAL TRIAL: NCT02766881
Title: Evaluation of the Ductal Carcinoma In Situ Score for Decisions on Radiotherapy in Patients With Low/Intermediate Risk DCIS
Brief Title: Evaluation of the DCIS Score for Decisions on Radiotherapy in Patients With Low/Intermediate Risk DCIS
Acronym: DUCHESS
Status: Completed | Type: Observational
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Other Study IDs: OCOG-2016-DUCHESS
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2019-08

CONDITIONS: DCIS
Keywords: Ductal Carcinoma in Situ; DSC; Breast Conserving Surgery
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — patient's tumour sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with DCIS: Whether patients with DCIS receive radiotherapy based on Oncotype DX DCIS score, radiation oncologist treatment recommendation and patient's decision.

SUMMARY:
To evaluate whether the use of the Oncotype DX DCIS score can guide delivery of radiation in women with low to moderate risk DCIS who have had breast conserving surgery

DETAILED DESCRIPTION:
A prospective cohort study, conducted in Canada, to evaluate whether the use of the DCIS score changes the treatment recommended and the treatment received in women with low to moderate risk DCIS following breast conserving surgery who are candidates for radiation therapy. We plan to study 280 eligible, consenting women who will have their tumour tissue specimen sent to Genomic Health to assess their DCIS score.

At each centre, all patients with DCIS referred to radiation oncology will be documented. When a physician identifies an eligible patient, the patient will be approached by the referring physician or delegate to voluntarily provide informed consent to participate in this study. Consenting patients will be registered through the Ontario Clinical Oncology Group's (OCOG) web-based registration system. Data related to the patient demographics, surgery details, and tumour characteristics will be collected. The preliminary treatment recommendation and patient preference for treatment will be documented. Patient Decisional Conflict will be documented by the patient using the Decisional Conflict Scale (DCS). The patient's tumour specimen will be sent for analysis to Genomic Health. DCIS score results will be sent to the referring physician. OCOG will also receive the DCIS score results. The final treatment recommendation, patient preference, and treatment received by the patient will be documented. Patient decisional conflict will be documented by the patient using the DCS. The study data will be verified by source documentation.

ELIGIBILITY:
Inclusion Criteria:

(1) Women with newly diagnosed breast cancer treated by definitive surgery with histological evidence limited to DCIS.

Exclusion Criteria:

1. Age < or = 45;
2. Treated by mastectomy;
3. Surgical margins of <1mm;(re-excisions may be performed where results are regarded as clear margins, these cases will not exclude patients);
4. Tumour size >2.5cm;
5. Any invasive breast cancer including micro invasion;
6. Histological evidence of multifocality (defined as having more than one distinct focus of DCIS with >5mm of intervening benign breast tissue in one quadrant of the breast);
7. Any associated lobular carcinoma in situ;
8. Previous diagnosis of ipsilateral invasive carcinoma or DCIS of the breast;
9. Any contraindication for whole breast irradiation such as chronic heart or lung disease or previous ipsilateral chest wall radiotherapy;
10. Physician/patient unwilling to comply with study protocol; and
11. Inability to provide informed consent (e.g. dementia or severe cognitive impairment).

Min Age: 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort study conducted in Ontario in women with a low to moderate risk DCIS following breast conserving surgery who are candidates for radiation. Eligibility status should be confirmed by the referring physician or delegate prior to enrollment. It is important that no exceptions are made to the eligibility criteria. Questions related to eligibility requirements and/or specific criteria should be addressed with OCOG prior to enrollment
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in radiotherapy treatment recommendation made by physician | 2.5 years
  The primary outcome is change in treatment recommendation by the radiation oncologist. Physicians will be asked to indicate their preliminary treatment recommendation at the first visit based on clinical factors alone. They will be asked to describe course of radiation including dose and number of fractions. They will then be asked to make a final treatment recommendation when the DCIS score is available. If the physician final recommendation is not consistent with the DCIS score predicted treatment, they will be asked to indicate reasons for their recommendation. If radiation is recommended, they will be asked to indicate the treatment prescription including dose and number of fractions. The actual treatment received by the patient will also be collected.

SECONDARY OUTCOMES:
Change in radiotherapy treatment preference by patient | 2.5 years
  Secondary outcomes will include change in treatment preference by the patient for radiotherapy and change in recommendations by the physician for hormonal therapy or further surgery. It will also compare physician's prediction of LR with or without radiation that is estimated by the DCIS score. Finally, change in level of patient decisional conflict as measured by DCS will also be collected. The DCS was developed and used to evaluate the effect of decision aids on decision making by health consumers.The assumption was that decision aids would reduce the uncertainty and confusion in choosing a course of action. Decisional conflict is a state of uncertainty about the course of action to take.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Rakovitch, M.D., Principal Investigator — Sunnybrook Health Sciences Odette Cancer Centre; Tim Whelan, M.D., Principal Investigator — Juravinski Cancer Centre
Locations (12):
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Vancouver Island, Victoria, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Genomic Health will provide results to referring physician, OCOG will have access to results

REFERENCES:
- See also: OCOG website accessed by clinical centres — http://www.ocog.ca